CLINICAL TRIAL: NCT07059169
Title: An Exploratory Clinical Study of the Safety, Tolerability, and Initial Efficacy of Targeted Cluster of Differentiation 19 (CD19) CAR-T Therapy for Refractory Autoimmune Diseases
Brief Title: CAR-T Therapy for Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LiangZou (Industry)
Responsible Party: Sponsor-Investigator, LiangZou, professor, Shenzhen Genocury Biotech Co., Ltd.
Organization: Shenzhen Genocury Biotech Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY CT-24-003
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-T for the treatment of refractory autoimmune diseases (Experimental): CD19 CAR-T for the Treatment of refractory autoimmune diseases subjects who meet the inclusion criteria will receive intravenous JY231 injection. JY231 injection infusion will produce CAR-T cells in the body.
  Interventions: Drug: JY231 (JY231 injection)

INTERVENTIONS:
Drug: JY231 (JY231 injection) — JY231 injection is administered intravenously and produces autologous CAR-T cells in the patient's body some time after infusion.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with refractory autoimmune diseases. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of CD19 CAR-T in the treatment of refractory autoimmune diseases.

DETAILED DESCRIPTION:
This open-label, single-arm study aims to evaluate the efficacy and safety of in vivo CAR-T cell therapy in patients with refractory autoimmune diseases. The study includes two pretreatment regimens: lymphodepletion and non-lymphodepletion.

Under the lymphodepletion regimen, after enrollment, patients will undergo leukapheresis followed by 3-5 days of fludarabine and cyclophosphamide lymphodepletion therapy. Subsequently, JY231 injection (CAR-T cell therapy) and autologous Peripheral blood mononuclear cell(PBMC) will be concurrently administered via double-lumen catheter intravenous infusion.

The non-lymphodepletion regimen involves direct infusion of JY231 injection without prior lymphodepletion.

Following infusion, subjects will undergo safety and efficacy assessments for up to 24 months to determine whether disease control is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, regardless of gender, signed with informed consent (ICF).
2. Diagnosed as one of the following diseases: Systemic lupus erythematosus (SLE)；Sjogren's syndrome (SS) ; Systemic Scleroderma (SSc); Dermatomyositis (DM); Anti neutrophil cytoplasmic antibody associated vasculitis (ANCA-AAV).
3. Patients who have been treated with ≥ 2 immunosuppressive agents for 3 months, or require ≥ 15mg glucocorticoids to maintain stable condition, or are intolerant to standard treatment, or have relative contraindications, and whose disease activity meets the following criteria:

   1. For SLE patients, SLEDAI ≥ 8 points;
   2. For SS patients, Sjogren's syndrome disease activity index(ESSDAI )≥ 14 points;
   3. For SSc patients, the modified skin score (mRSS) score ranges from 10 to 35 (including cutoff values) and is associated with interstitial pneumonia (ILD);
   4. For DM patients, diagnosed for at least 1 year;
   5. For ANCA-AAV patients, Birmingham Vasculitis Activity Score(BVAS) score ≥ 15 and ANCA antibodies.
4. Eastern Cooperative Oncology Group(ECOG) 0-1 points;
5. The evaluation of important organ functions meets the following conditions:

   1. Blood count: hemoglobin ≥ 60g/L, platelet count ≥ 30 × 109/L;
   2. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 55%, no significant abnormalities observed on electrocardiogram;
   3. Renal function: estimated glomerular filtration rate(eGFR) ≥ 30 mL/min/1.73m2;
   4. Liver function: Aspartate Aminotransferase(AST) and Alanine Transaminase(ALT) ≤ 3.0 upper limit of normal(ULN), total bilirubin ≤ 2.0 ULN;
   5. Pulmonary function: diffusion capacity of the lung for carbon monoxide(DLCO) ≥ 40% expected value; forced vital capacity(FVC) ≥ 50% of expected value;
   6. Having single or intravenous blood collection standards and no other contraindications for cell collection;
6. The urine pregnancy test results of subjects of childbearing age are negative, and they agree to take effective contraceptive measures during the trial period, until one year after infusion;
7. The patient or their guardian agrees to participate in this clinical trial and signs an informed consent form, indicating their understanding of the purpose and procedures of this clinical trial and willingness to participate in the study.

Exclusion Criteria:

1. Previously received Chimeric Antigen Receptor T cell(CAR-T) therapy;
2. Suffering from severe diseases of the heart, liver, lungs, blood system, and endocrine system, the researcher has determined that the risk of participating in the trial is higher than the benefit;
3. Active or uncontrollable infections that require systemic treatment within the first week of screening;
4. Previously received hematopoietic stem cell transplantation or solid organ transplantation (excluding corneal and hair transplantation), or screened for acute graft-versus-host disease (GVHD) with grade 2 or above in the first two weeks;
5. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive and the hepatitis B virus(HBV) DNA titer in peripheral blood is greater than the normal reference value; Or hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA titer detection greater than the normal reference range; Or positive for human immunodeficiency virus (HIV) antibodies; Or those who test positive for syphilis; Or positive for cytomegalovirus (CMV) DNA detection;
6. Received live vaccine within 4 weeks prior to screening;
7. Pregnancy test positive individuals;
8. Patients with malignant tumors and other malignant diseases before screening, in addition to fully treated cervical cancer in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
9. Screening patients who have participated in other clinical trials within the first three months;
10. Other researchers believe that it is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan No.1 Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No